CLINICAL TRIAL: NCT06403163
Title: Biological Transfusion Efficiency Registry Transfusion Surveillance in Anaesthesia
Brief Title: Transfusion Surveillance in Anaesthesia
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STAR
Record Dates: First submitted 2022-02-08; First posted 2024-05-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Transfusion Reaction; Transfusion Related Complication; Anesthesia; Anesthesia; Shock; Side Effect; Fresh Blood Stool; Blood Coagulation Disorder; Blood Loss
Keywords: transfusion; monitoring; emergency situation; shock; fresh frozen plasma
MeSH Terms: conditions — Transfusion Reaction; Shock; Gastrointestinal Hemorrhage; Blood Coagulation Disorders; Hemorrhage; Emergencies | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transfused patients: patients who received an hemostatic product
  Interventions: Procedure: Transfusion

INTERVENTIONS:
Procedure: Transfusion — Transfusion of an hemostatic product

SUMMARY:
the aim of this register is to collect exhaustively the different data available surrounding a transfusion act in the context of an active haemorrhage. The aim is to allow different modelling and analysis related to emergency transfusion.

DETAILED DESCRIPTION:
the aim of this register is to collect exhaustively the different data available surrounding a transfusion act in the context of an active haemorrhage. The aim is to allow different modelling and analysis related to emergency transfusion.

Patients will be informed at the time of the anaesthesia consultation about the inclusion in the registry.

The data will be collected from the patients' files by the investigators of the centre without modifying their management.

The data collection period will not exceed the period of acute management.

ELIGIBILITY:
Inclusion Criteria:

* all patients who have received an hemostasis product

Exclusion Criteria:

* patient who refused to consent to data analysis and study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient who received an hemostasis product during an hemorrhagic situation
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemostatic evolution through transfusion event | 12 hours
  evolution of APTT (seconds)
ROTEM measures evolution through transfusion event | 12 hours
  evolution of APTEMCT (seconds)
Haematologic measures evolution through transfusion event | 12 hours
  evolution of hemoglobin (g/dL)
ionic measures evolution through transfusion event | 12 hours
  evolution of lactate (mmol/L)

SECONDARY OUTCOMES:
Mortality at one month | one month
  Mortality at one month

CONTACTS AND LOCATIONS:
Locations (1):
- Université libre de Bruxelles, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No